CLINICAL TRIAL: NCT01730963
Title: Multi-Reader Multi-Case Study to Identify Uterine Contractions Recorded From Laboring and Nonlaboring Patients by Practicing Clinicians
Status: Completed | Type: Observational
Sponsor: Reproductive Research Technologies, LP (Industry)
Responsible Party: Sponsor
Other Study IDs: RRT-12-01
Record Dates: First submitted 2012-11-15; First posted 2012-11-21 (Estimated); Last update posted 2012-11-22 (Estimated); Status verified 2012-11

CONDITIONS: Pregnancy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Pregnant, Preterm, In Labor: Gestation Age at or less than 36 weeks, clinically determined to be in labor
- Pregnant, Preterm, Nonlaboring: Gestation Age at or less than 36 weeks, clinically determined to not be in labor
- Pregnant, Term, Nonlaboring: Gestation Age more than 36 weeks, clinically determined to not be in labor

SUMMARY:
This multi-reader multi-case study was designed to evaluate the performance of SureCALL® Labor Monitor® (SureCALL®) directly to the standard Tocodynamometer device (TOCO).

DETAILED DESCRIPTION:
The SureCALL® Labor Monitor® (SureCALL®) is a transabdominal electromyography monitor intended to measure uterine activity. It is intended for use on pregnant women, with singleton pregnancies, using surface electrodes on the maternal abdomen. The device is intended for use by healthcare professionals in a clinical setting.

This multi-reader multi-case study was designed to evaluate the performance of SureCALL® to the predicate Tocodynamometer device (TOCO).

This study involved 25 women at a Gestational Age of 36 weeks or less and 5 women at a Gestation Age of greater than 36 and not in labor at five clinical sites. Each study subject was instrumented with two technologies for measuring uterine activity:

1. Standard tocodynamometer attached to the maternal abdomen,
2. SureCALL® with a set of abdominal surface electrodes for uterine electromyography attached to the maternal abdomen

An assessment was obtained and quantified from masked, qualified clinical obstetrician readers for the evaluation of the equivalence of both labor monitor devices by identifying in isolation the individual uterine contraction signals and the peak of each contraction signal as recorded by each labor monitor device.

ELIGIBILITY:
Inclusion Criteria:

* Singleton Pregnancy
* Informed Consent Required

Exclusion Criteria:

* Multifetal Pregnancy
* Informed Consent Not Given

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women with uncomplicated singleton pregnancies
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2007-01; Primary Completion 2011-12 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Comparison of SureCALL® and Tocodynamometer Detection of Contraction Events, as Identified by Readers | 9 - 41 Minutes
  Agreement will be assessed by coefficient of individual agreement (CIA) derived from a dataset of all Reader-marked contractions. In addition, sensitivity and false positive rate per hours will be estimated for each patient by each reader. If CIA ≥ 0.445 (Barnhart, 2007, section 3) or CIA>0.8, Pan 2010), the SureCALL® is not significantly different than the TOCO.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy B Waterhouse, MD, Study Director — Reproductive Research Technologies, LP
Locations (5):
- United States (5):
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - Southeast Texas OB/GYN Associates, Beaumont, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Woman's Hospital of Texas, Houston, Texas